CLINICAL TRIAL: NCT01082484
Title: Cutaneous Iontophoresis of Iloprost and Treprostinil in Healthy Volunteers
Acronym: INFLUX-IT-VS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-016301-42
Record Dates: First submitted 2010-02-09; First posted 2010-03-08 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: Healthy volunteers; iontophoresis
MeSH Terms: interventions — treprostinil; Iloprost; Sodium Chloride

ARMS (3):
- Treprostinil (Experimental): Treprostinil iontophoresis (250, 25 and 2.5 microM)
  Interventions: Drug: treprostinil
- Iloprost (Experimental): Iloprost iontophoresis (200, 20 and 2 microM)
  Interventions: Drug: iloprost
- NaCl 0.9% (Placebo Comparator)
  Interventions: Drug: NaCl 0.9%

INTERVENTIONS:
Drug: treprostinil — Cutaneous iontophoresis at 20 microA/ 100 microA during 20 min
  Arms: Treprostinil
Drug: iloprost — Cutaneous iontophoresis at 20 microA/ 100 microA during 20 min
  Arms: Iloprost
Drug: NaCl 0.9% — Cutaneous iontophoresis at 20 microA/ 100 microA during 20 min
  Arms: NaCl 0.9%

SUMMARY:
The purpose of this study is to test whether prostacyclin analogues' cathodal iontophoresis induce a cutaneous vasodilation in healthy volunteers's forearm, without local side effects.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* age above 18

Exclusion Criteria:

* any chronic disease
* any drug intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Amplitude of forearm cutaneous vasodilatation assessed using laser Doppler imaging | 24 hours

SECONDARY OUTCOMES:
Local tolerance assessed clinically | Day 0 and after 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Unité de Pharmacologie Clinique, Inserm CIC3, CHU Grenoble, Grenoble, France

REFERENCES:
- [Derived] Blaise S, Roustit M, Hellmann M, Millet C, Cracowski JL. Cathodal iontophoresis of treprostinil induces a sustained increase in cutaneous blood flux in healthy volunteers. J Clin Pharmacol. 2013 Jan;53(1):58-66. doi: 10.1177/0091270011434352. Epub 2013 Jan 24. PMID 23400744